CLINICAL TRIAL: NCT00050206
Title: Olanzapine Versus Placebo in the Treatment of Mania in Adolescents With Bipolar I Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4360; F1D-MC-HGIU
Record Dates: First submitted 2002-11-26; First posted 2002-11-27 (Estimated); Last update posted 2007-06-12 (Estimated); Status verified 2007-06

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Olanzapine

INTERVENTIONS:
Drug: Olanzapine
Drug: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy (how well the drug works), safety, and any side effects of olanzapine compared to placebo in the treatment of mania in bipolar disorder in adolescents. Both the potential benefits and side effects of olanzapine will be evaluated throughout this trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 13 to 17 years of age who must not yet have reached their 18th birthday prior to Visit 1, when informed consent is obtained.
* Patients must have a diagnosis of bipolar I disorder and currently display an acute mania or mixed episode.
* Both the patient and the patient's parent/authorized legal representative must understand the nature of the study and must sign a document granting consent.
* Female patients of child-bearing potential must test negative for pregnancy at the time of enrollment based on a serum pregnancy test.

Exclusion Criteria:

* Female patients who are either pregnant or nursing.
* Current diagnosis of schizophrenia, schizophreniform disorder, or schizoaffective disorder.
* Patient with acute or unstable medical conditions, such that intensive care unit hospitalization for the disease is anticipated within 6 months.
* Patients who have previously not responded to an adequate dose and/or duration of olanzapine treatment.
* Patients who have been judged clinically to be serious suicidal risks.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130
Dates: Start 2002-11; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of a flexible dose of olanzapine compared with placebo in the treatment of mania in bipolar I disorder (manic or mixed episode associated with bipolar I disorder, with or without psychotic features) in adolescents

SECONDARY OUTCOMES:
Assess additional efficacy as measured by Y-MRS,CGI-BP Severity of Illness, CGI-BP Severity of Illness (CGI-BP Severity of Mania, CGI-BP Severity of Depression, and CGI-BP Severity Overall)
Assess additional efficacy as measured by Children's Depression Rating Scale-Revised (CDRS- R);Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version: Investigator Administered and Scored (ADHDRS-IVPI) and Overt Aggression Scale (OAS).
Assess the safety of olanzapine and quality of life associated with olanzapine compared with placebo.
Compare the frequency of response of up to 3-weeks, double-blind treatment and up to an additional 26 weeks of open-label olanzapine treatment

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Xiao L, Ganocy SJ, Findling RL, Chang K, DelBello MP, Kane JM, Tohen M, Xiang YT, Correll CU. Baseline Characteristics and Early Response at Week 1 Predict Treatment Outcome in Adolescents With Bipolar Manic or Mixed Episode Treated With Olanzapine: Results From a 3-Week, Randomized, Placebo-Controlled Trial. J Clin Psychiatry. 2017 Nov/Dec;78(9):e1158-e1166. doi: 10.4088/JCP.16m10923. PMID 28922591
- [Derived] Kryzhanovskaya LA, Robertson-Plouch CK, Xu W, Carlson JL, Merida KM, Dittmann RW. The safety of olanzapine in adolescents with schizophrenia or bipolar I disorder: a pooled analysis of 4 clinical trials. J Clin Psychiatry. 2009 Feb;70(2):247-58. doi: 10.4088/jcp.08m03538. Epub 2009 Feb 10. PMID 19210948
- [Derived] Tohen M, Kryzhanovskaya L, Carlson G, Delbello M, Wozniak J, Kowatch R, Wagner K, Findling R, Lin D, Robertson-Plouch C, Xu W, Dittmann RW, Biederman J. Olanzapine versus placebo in the treatment of adolescents with bipolar mania. Am J Psychiatry. 2007 Oct;164(10):1547-56. doi: 10.1176/appi.ajp.2007.06111932. PMID 17898346
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com